CLINICAL TRIAL: NCT04748185
Title: Immunogenicity and Safety of Commercially Available Vaccines Against Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) in Patients With Hematologic Malignancies and Associated Precursor Conditions
Brief Title: Immunogenicity and Safety of Commercially Available Vaccines Against SARS-CoV-2 (COVID-19) in Patients With Hematologic Malignancies
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20-012589
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Monoclonal B-Cell Lymphocytosis; Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; B-cell Non Hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: Lymphoma; Covid-19 Vaccine; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Hodgkin Disease; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
D1. Primary Objective:

1. Determine the immunogenicity of FDA approved COVID-19 vaccination in patients with hematologic malignancies

D2. Secondary Objectives:

1. Assess the safety of FDA approved COVID-19 vaccination in patients with hematologic malignancies
2. Analyze the kinetics of immunogenic response over time after receipt of the COVID-19 vaccination
3. Compare the immunogenicity of different COVID-19 vaccinations that will be approved by the FDA
4. Analyze advanced flow immunophenotyping of innate and adaptive immune blood cells in all participants and correlate with response to vaccination

ELIGIBILITY:
Inclusion Criteria:

1. Patients must not have received any prior COVID-19 vaccination
2. Patients must have any one of the following diagnosis:

   a. Monoclonal B-cell lymphocytosis b. Chronic lymphocytic leukemia/small lymphocytic lymphoma c. B-cell Non-Hodgkin's lymphoma: i. Follicular lymphoma ii. Mantle cell lymphoma iii. Diffuse large B-cell lymphoma iv. Marginal zone lymphoma v. Burkitt lymphoma vi. Double hit/triple hit lymphoma vii. Lymphoplasmacytic lymphoma/Waldenstrom's macroglobulinemia d. Hodgkin lymphoma

Exclusion Criteria:

1. Receipt of any vaccination (e.g., influenza, recombinant zoster) 2 weeks prior to registration
2. Prior chemotherapy, immunotherapy or oral agent therapy that was completed >12 months prior to enrollment. NOTE: patients who are on oral agents for the treatment of their underlying malignancy will be allowed. Some of these medication classes include Bruton tyrosine kinase inhibitor (BTKi), BCL2 antagonists, PI3 kinase inhibitors, immunomodulatory agents, among others. Please contact the Principal Investigator for any clarification about these medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will submit peripheral blood samples a) prior to first dose of vaccination; b) prior to receipt of the second dose of vaccination; c) 14 days following the second dose; and d) 3, 6 and 12 months following the first dose of the vaccination. For patients at time points a, b, and c blood samples can be collected up to 3 days prior; and at time point d +/- 10 days.
  Patients who are seen at Mayo Clinic in Rochester, MN can collect their blood through a venipuncture at the clinic. For patients who are to receive vaccination locally, a blood kit will be mailed for the patients to get research bloods collected and sent to Mayo Clinic.
  All patients will also complete a diary of adverse reactions (Appendix I) daily for 7 days after receipt of each dose of the vaccine. Patients will be asked to contact their primary care provider or hematologist if they have any side effects from the vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Humoral Immunogenicity | Assessed 14 days following the second dose of the vaccine
  Number of participants who have detectable antibodies to SARS-Co-V2 vaccination
Cellular Immunogenicity | Assessed 14 days following the second dose of the vaccine
  Number of participants who have a SARS-CoV-2 specific memory B cell ELISPOT response
Cellular Immunogenicity | Assessed 14 days following the second dose of the vaccine
  Number of participants who have a SARS-CoV-2 specific IFNγ ELISPOT T cell response

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Parikh, M.B.B.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials